CLINICAL TRIAL: NCT01927432
Title: Ultrasound Characterization of Ovarian Follicle Dynamics in Women With Amenorrhea
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB #: 0908000633
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Oligomenorrhea; Amenorrhea; Polycystic Ovary Syndrome (PCOS)
Keywords: Polycystic Ovary Syndrome (PCOS); Nutrition; Metabolism; Antral follicle growth; Menstrual Cyclicity
MeSH Terms: conditions — Oligomenorrhea; Amenorrhea; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum, subcutaneous fat
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Regular menstrual cycles: Adult women will be assigned to this category if they report a history of regular menstrual cycles.
- Irregular menstrual cycles: Adult women will be assigned to this category if they report a history of irregular menstrual cycles, including women with a pre-existing diagnosis of PCOS.

SUMMARY:
In women with regular menstrual cycles, antral follicles have been shown to grow in synchronous cohorts, called waves, 2-3 times in a menstrual cycle. It is unknown whether these waves of follicle growth also occur in women with amenorrhea or if there is abnormal/absent follicle growth. Further, oligo- or amenorrhea has been associated with metabolic disturbances, such as over- or under-nutrition, central obesity and insulin resistance. Yet, mechanisms whereby metabolic factors influence folliculogenesis in women are poorly understood. To understand potential mechanisms, the investigators plan to characterize follicle growth dynamics in women with or without regular menstrual cycles and identifying key metabolic differences in these women which may be important in normal follicle development and fertility.

DETAILED DESCRIPTION:
In the ovaries, eggs rest in fluid filled sacs called follicles. When follicles grow they form small fluid-filled cysts that can be easily seen when we use ultrasound to view the ovaries. In women with regular menstrual cycles, groups of 10 to 20 follicles grow and regress at 2 or 3 different times during their cycle (usually over a 28- day period). Several of these follicles grow to a stage where they begin to develop the potential to ovulate - but in general only one follicle is chosen to ovulate. Thus, at any given time during the menstrual cycle, numerous fluid-filled follicles can be visualized in a woman's ovaries at various stages of development using transvaginal ultrasonography. In women with absent or infrequent menstrual cycles, very little is known about the growth patterns of their follicles and how factors such as metabolic hormones, might play a role in the failure to ovulate. Being underweight or overweight increases your chances of having irregular or absent menstrual cycles and that a history of abnormal reproductive function compounds a woman's risk for chronic diseases such as infertility, diabetes, hypertension, atherosclerosis and certain cancers. This is particularly the case for women with polycystic ovary syndrome (PCOS) that have menstrual cycles that appear to worsen or improve depending on their body weight and metabolic status. PCOS is an endocrine disorder that affects 6-12% of reproductive-aged women within the general population. The hallmark features of PCOS are menstrual irregularity, increased levels of androgens, and polycystic ovaries. The current diagnostic criteria require 2 out of 3 of these features to be present for the diagnosis, therefore a number of phenotypes of PCOS exist. However, the metabolic and reproductive differences across the phenotypic spectrum of PCOS are not well understood. Women with PCOS characteristically have polycystic ovaries, where up to 10 times more follicles are present in the ovary at any given time. Further, the follicle-size populations and overall distribution throughout the ovary varies in women - follicles may be situated around the periphery of the ovary or may be distributed throughout the ovary. Presumably these small follicles are arrested in development - but emerging data from the Lujan laboratory suggest that this is not the case. It is assumed that ovulation does not occur and that follicles do not grow in a normal wave pattern. In truth, no study has ever looked to see whether follicles are actually growing, regressing or are arrested in women with irregular/absent menstrual cycles. By comparing follicle wave dynamics, reproductive hormones and markers of metabolism in women with regular and irregular menstrual cycles, the researchers plan to identify what factors might explain why fertility potential and long-term health are compromised in some women but not in others. Further, we will determine if any of these metabolic factors are unique to PCOS representing specific metabolic risks or follicle growth impairment. The ultimate goal of this research is to understand how body composition, nutrition and metabolism regulate follicle development in women so we can better develop lifestyle and drug therapies to help women preserve their fertility and long-term health. Since obesity has recently become the leading cause of infertility in North America, these studies are especially important.

To accomplish our objective, the investigators plan to recruit up to 40 women with regular menstrual cycles and up to 40 women with irregular/absent menstrual cycles. Our goal is to recruit an equal number of women in each group such that they are matched for age (18 - 35 years old) and body mass index (BMI; Normal weight = 18 - 24 kg/m2; Overweight = 25 - 29 kg/m2; Obese = 30kg/m2). Women will undergo serial ultrasonographic of their ovaries every other day from ovulation to ovulation in women with regular menstrual cycles or for 5 weeks in women with cycle irregularity. Blood samples will be collected at each visit. Ultrasound scans of the ovaries will be assessed for the total number, size, and distribution of follicles using ultrasound imaging techniques. Blood samples collected will be assayed to determine serum concentrations of luteinizing hormone (LH), follicle stimulating hormone (FSH), estradiol, progesterone, anti-müllerian hormone (AMH), and inhibin B. During day 3-5 in women with regular menstrual cycles or at a time where no dominant follicle or corpus luteum is present, an early morning visit will be conducted to assess the following metabolic parameters : (1) 75-gram oral glucose tolerance test to characterize glucose and insulin dynamics at 0, 30, 60, 90, and 120 minutes post-glucose ingestion; (2) dual X-ray absorptiometry (DXA) scan to quantify body fat and lean muscle distribution; (3) vitals and anthropometry assessment to measure waist and hip circumference, height, weight, blood pressure, and heart rate, and (4) fasting blood tests to detect serum concentrations of androgens (i.e., total testosterone, androstenedione, free androgen index) and serum markers of metabolic syndrome (i.e., lipids and hemoglobin A1C); (5) optional subcutaneous fat biopsy to analyze fat cells, which represent a site of reproductive hormone synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 35 years
* BMI ≥ 18 kg/m2
* If ≥ 21 years old, must have had healthy pelvic exam w/in past 2 years

Either:

* Regular menstrual cycles (21-35 days);
* Irregular menstrual cycles (>36 days) with or without a previous diagnosis of PCOS from a primary care provider

Exclusion Criteria:

* Current use of medication(s) known or suspected to interfere with reproductive function (eg. oral contraceptives) or insulin sensitivity
* Pregnant or breastfeeding
* Not otherwise healthy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women must be able to transport to Cornell University in Ithaca, NY. Eligible participants are between 18-35 years with a BMI of 18 kg/m2 or higher. Women are screened and enrolled following consent based on their response to our advertisements. Enrollment is restricted to the geographical area.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2011-09; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Follicle number | 4-5 weeks
  The number of all antral follicles in each ovary will be determined using ultrasonography for each participant. Changes in follicle number over time will be compared between groups.
Follicle diameter | 4-5 weeks
  The diameter of all follicles >2mm will be determined using ultrasonography for each participant. Changes in follicle diameter over time will be compared between groups.

SECONDARY OUTCOMES:
Ovarian Volume | 4-5 weeks
  The size of each ovary will be determined using ultrasonography for each participant during study participation and compared between groups.
Anti-Müllerian hormone | 4-5 weeks
  The serum AMH concentration will be determined during study participation and assessed in association with the change in follicle number, diameter and between groups.
Serum FSH concentration | 4-5 weeks
  The serum FSH concentration will be determined during study participation and assessed in association with the change in follicle number, diameter and between groups.
Serum LH concentration | 4-5 weeks
  The serum FSH concentration will be determined during study participation and assessed in association with the change in follicle number, diameter and between groups.
Serum progesterone concentration | 4-5 weeks
  The serum progesterone concentration will be determined during study participation, assessed in association with luteal dynamics and compared between groups.
LH-FSH ratio | 4-5 weeks
  The ratio of circulating LH to FSH concentrations will be determined for each participant and compared between groups.
Insulin sensitivity | 1 day
  Insulin sensitivity will be determined by administration of an oral glucose tolerance test and compared between groups.
Androgen concentrations | 1 day
  Total testosterone, androstenedione and free androgen index concentrations in serum will be determined and compared between groups.
Menstrual Cycle Length | 4-5 weeks
  Average menstrual cycle length as determined by self-reported history and the menstrual cycle length during study participation will be determined and compared between groups.
Hirsutism | 1 day
  Degree of hirsutism as judged by the Ferriman-Gallwey scale will be determined and compared between groups.
Serum markers of metabolic syndrome | 1 day
  Lipids, glucose and HbA1C concentrations will be determined and compared between groups.
Blood Pressure | 1 day
  Blood pressure will be determined and compared between groups.
Body mass index | 1 day
  The ratio of weight to height will be determined and compared between groups.
Waist-to-hip ratio | 1 day
  The ratio of waist circumference to hip circumference will be determined and compared between groups.
Body fat distribution | 1 day
  Percentage and distribution of fat and lean mass as assessed using DXA technology will be compared between groups.
Subcutaneous fat biopsy (optional) | 1 day
  Fat cells, representing an important site of reproductive hormone production, will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Marla E. Lujan, PhD, Principal Investigator — Cornell University
Locations (1):
- Human Metabolic Research Unit, Cornell University, Ithaca, New York, United States

REFERENCES:
- [Derived] Oldfield AL, Carter FE, Reeves RE, Jarrett BY, Vanden Brink H, Lujan ME. Impact of a hypocaloric dietary intervention on antral follicle dynamics in eumenorrheic women with obesity. Hum Reprod. 2024 Apr 3;39(4):801-811. doi: 10.1093/humrep/deae017. PMID 38335228
- [Derived] Oldfield AL, Vanden Brink H, Carter FE, Jarrett BY, Lujan ME. Obesity is associated with alterations in antral follicle dynamics in eumenorrheic women. Hum Reprod. 2023 Mar 1;38(3):459-470. doi: 10.1093/humrep/dead007. PMID 36708012